CLINICAL TRIAL: NCT02749877
Title: Efficacy of Cognitive and Physical Trainings in Pediatric Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 196/15
Record Dates: First submitted 2016-04-12; First posted 2016-04-25 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Pediatric Cancer
Keywords: Pediatric Cancer; Training; Working Memory; Physical Activity; Brain Tumor; Physical Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity; Brain Neoplasms | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Training (Experimental): This group will undergo a working memory training program (Training A). The children will receive individual memory training based on the computer program Cogmed RM and will be supervised by trained neuropsychologists. Its efficacy in the use with children with cancer has been recently published. The children will undergo 25 training sessions "online"; each session takes about 45 minutes and consists of a selection of various tasks that target the different aspects of working memory.
  Interventions: Behavioral: Working Memory Training
- Physical Training (Experimental): This group will receive a physical training that can be executed at home (Training B). The training will be based on xbox Kinect games and comprise games and activities such as jump'n'run games, physical training, and dance activities. One training session will last approximately 45 minutes and will be performed 3 days a week over a period of 8 weeks (in total 25 sessions).
  Interventions: Behavioral: Physical Training
- Waiting Control Group (Active Comparator): This group will serve as a waiting control group and will receive either the physical or the working memory training program after completion of the Neuropsychological Assessment II
  Interventions: Behavioral: Working Memory Training; Behavioral: Physical Training

INTERVENTIONS:
Behavioral: Working Memory Training — (Training Details already described above)
  Arms: Cognitive Training; Waiting Control Group
Behavioral: Physical Training — (Training Details already described above)
  Arms: Physical Training; Waiting Control Group

SUMMARY:
Cancer survival comes at a price: pediatric cancer survivors have a high risk for a wide range of cognitive difficulties, particularly survivors of cancer involving the central nervous system (CNS, e.g., brain tumors [BT]) are prone to neurocognitive impairments in areas such as executive functions, working memory, attention, memory, visuospatial and motor skills, processing speed as well as language. The aim of this interdisciplinary longitudinal study is to extend empirical knowledge on training and transfer effects in children with a history of cancer. It is hypothesized that early cognitive and physical interventions affect the remediation of pediatric cancer survivors in terms of cognitive functions. These changes are further hypothesized to be associated with white matter changes.

DETAILED DESCRIPTION:
Aims and Hypotheses:

The overall purpose of this study is threefold: first, this study aims to deepen the knowledge about particular patterns of long-term cognitive impairment in pediatric cancer survivors. Understanding the nature of cognitive deficits in this population will be helpful for developing tailored therapeutic strategies. Second, the availability of well-designed child-friendly evidence-based training is of major clinical relevance to prevent school problems and further decline of cognitive functions. Third, the detection of training-induced neuronal changes in white-matter structure will give insight into the functional plasticity of the child's brain. In addition, training-induced changes in white matter would build strong evidence for the effect of the particular intervention.

The following hypotheses will be assessed in particular in the present study:

1. Children with history of brain tumors (BT) show particular problems in memory and attention, resulting in a general deficit in several cognitive areas. Children with a history of cancer without involvement of the CNS show fewer problems than children with a history of cancer with BT in the same cognitive domains but more problems than healthy control children.
2. Standardized working memory training leads to improvement of working memory performance. Transfer of the training effect especially to the areas of executive functions, memory and attention is expected.
3. Physical training leads to improvement of coordination, endurance and motor strength. A transfer to several cognitive areas (i.e. executive functions) and physical self-concept is expected.
4. After working memory training and physical training, the white matter structure of the patients will show significant changes in fractional anisotropy. There will also be changes in functional connectivity.
5. Neuropsychological effects of training will still be present after 6 months post training for both experimental groups.

All comparisons will be carried out on an individual level (intra-individual level, primary objective) as well as on an inter-individual level (between-groups comparisons, secondary objective). The level of significance is set to α = 0.05.

Participants:

Cancer Survivors: Researchers will include 150 children and adolescents aged 7-16 years who received an initial diagnosis of cancer with / without CNS (central nervous system) involvement in the past 10 years and terminated their treatment (surgery, radiation, and / or chemotherapy) at least 12 months prior to their participation in the study. Cancer survivors will be recruited at two different specialized pediatric units in Switzerland. In order to minimize the heterogeneity of the sample, children with a history of cancer without CNS involvement and only surgical removal of the tumor without subsequent radiation and / or chemotherapy will be excluded from the study. Because of the increased likelihood of drop-out of children with a history of cancer in a longitudinal study, more than the statistically required quantity of participants (> 25 children per group) will be recruited to reach sufficient statistical power.

Healthy Controls: 40 healthy children and adolescents (matched for age and gender) will be included in the first assessment and serve as a healthy control sample. They will be recruited mainly via their siblings, who are included in the cancer survivor group and also from personal acquaintances among hospital staff and the study collaborators.

Design The present study is designed as a randomized stratified controlled trial including two intervention groups, one waiting group (children with a history of cancer [both CNS+ and CNS-] and a healthy control group (matched for age and gender). Some children of the patient group will be allocated to a waiting-control group to determine the training effects (their training starts later on). After random assignment to the respective conditions, the interventional material (XBOX or computer), will be installed at the participants home. Thereby, a supervised first training session will take place. The executive functions before and after as well as more details on the effects of a single intervention session (on enjoyment, arousal etc.) will be examined. Subsequently, the respective group will either follow a standardized, computerized working memory training or a physical training. Neuropsychological assessment will be carried out before the intervention / training and re-performed with all participants at the end of the memory training or physical training and at 6 months posttraining. Structural and functional imaging will be performed prior and shortly after working memory training and physical training. A 3 Tesla whole body MRI system will be used (Siemens; Erlangen, Germany). Anatomical imaging will be obtained using a sequence for T1 weighted structural brain imaging with whole brain coverage. Structural connectivity images will be acquired by using a q-ball sequence, functional connectivity will be measured by using a multiband echo planar imaging sequence (MB EPI). Pre- and post-processing of the structural data will be performed using SPM8 (Welcome Departement of Imaging Neuroscience, London) and MATLAB programs (MATLAB version 8.2). In order to perform functional connectivity analyses, the CONN fMRI connectivity toolbox 13.1 (Whitfield-Gabrieli & Nieto-Castanon, 2012) is used. The fractional anisotropy maps are provide by the Siemens software and can be directly used for further statistical evaluation.

Interventions:

All 150 participants with a history of cancer will be randomly but in a stratified manner assigned to 3 groups (group A, B and C) (see Fig.1).

Training A: Group A (n1= 25 CNS+, n2 = 25 CNS-) will undergo working memory training program. The children will receive individual memory training based on the computer program Cogmed RM (Klingberg et al., 2005) and will be supervised by trained neuropsychologists. Its efficacy in the use with children with cancer has been recently published (e.g. Hardy et al., 2012). The children will undergo 25 training sessions "online"; each session takes about 45 minutes and consists of a selection of various tasks that target the different aspects of working memory. The difficulty level of the training is always adjusted based on the user's performance. The children will perform the memory training program at home over a period of 8 weeks. The child and a licensed Cogmed RM coach (neuropsychologist) will review and monitor the results of each day's training online. In an initial session at the Hospital (Zurich or Bern) the Cogmed RM coach plans and structures the training together with the child and the parents. The coach will provide weekly supervision and feedback on the child's performance and progress via phone call to the child's home. In the closing session with the child and the parents, the training experience will be reviewed .

Training B: Group B (n1= 25 CNS+, n2 = 25 CNS-) will receive a physical training that can be executed at home. The training will be based on xbox Kinect games (e.g. Shape Up) and comprise games and activities such as jump'n'run games, physical training, and dance activities. All material will be provided by the Inselspital Bern. One training session will last approximately 45 minutes and will be performed 3days a week over a period of 8 weeks.

Group C (n1= 25 CNS+, n2 = 25 CNS-) will serve as a waiting control group and will receive either the physical or the working memory training program after completion of the Neuropsychological Assessment II.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature of participants and / or parents / legal guardians
* Age 7-16 years
* A history of cancer either with or without CNS involvement in the past 10 years and termination of treatment at least 12 months prior to participation in the study
* Treatment of cancer including either radiation and / or chemotherapy in addition to surgical tumor removal if the cancer did not involve the CNS

Exclusion Criteria:

* Contraindication to cognitive training and / or presentation of physical activity on a TV- or computer screen, in particular epilepsy
* Any other instable neurological or physical condition
* Cancer treatment of only surgical intervention without subsequent radiation and / or chemotherapy if the CNS was not affected
* For female participants: Pregnancy or breast feeding; or, intention to become pregnant during the course of the experiment; or, lack of safe contraception (defined as: female participants of childbearing potential, not using a medically reliable method of contraception, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases). A pregnancy test will be provided for participants of ages 14 and older
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2017-01; Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Participant's individual score in executive functions (Subtest Block Recall; Color-Word Interference Test) | baseline - 8 weeks - 3 months
  The primary endpoint in this study will be the participant's scores in executive functions based on the model of Miyake et al. (2000) which will be assessed using two different subtests: The subtest Block Recall from the Working Memory Test Battery for Children, WMTB-C (Pickering & Gathercole, 2001) and the Color-Word Interference Test from the Delis-Kaplan Executive Function System™ (D-KEFS™, (Delis, Kaplan, & Kramer, 2001).These tests will be administered at each neuropsychological testing, specifically, before and after the training intervention. It is expected to find a statistically significant amelioration in performance after the intervention (effect size f = 0.14 at a level of significance of α =0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Leibundgut, MD Prof, Principal Investigator — Inselspital Bern, Switzerland
Locations (1):
- University Children's Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Benzing V, Spitzhuttl J, Siegwart V, Schmid J, Grotzer M, Heinks T, Roebers CM, Steinlin M, Leibundgut K, Schmidt M, Everts R. Effects of Cognitive Training and Exergaming in Pediatric Cancer Survivors-A Randomized Clinical Trial. Med Sci Sports Exerc. 2020 Nov;52(11):2293-2302. doi: 10.1249/MSS.0000000000002386. PMID 33064404
- [Derived] Benzing V, Eggenberger N, Spitzhuttl J, Siegwart V, Pastore-Wapp M, Kiefer C, Slavova N, Grotzer M, Heinks T, Schmidt M, Conzelmann A, Steinlin M, Everts R, Leibundgut K. The Brainfit study: efficacy of cognitive training and exergaming in pediatric cancer survivors - a randomized controlled trial. BMC Cancer. 2018 Jan 3;18(1):18. doi: 10.1186/s12885-017-3933-x. PMID 29298678